CLINICAL TRIAL: NCT00768430
Title: Optimization of Intravenous Ketamine for Treatment-Resistant Depression: A Randomized, Placebo-Controlled, Triple-masked, Clinical Trial
Brief Title: Optimization of IV Ketamine for Treatment Resistant Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Sanjay Johan Mathew, MD, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GCO 07-0114
Record Dates: First submitted 2008-10-07; First posted 2008-10-08 (Estimated); Results first posted 2014-01-31 (Estimated); Last update posted 2014-01-31 (Estimated); Status verified 2013-12

CONDITIONS: Major Depressive Disorder (MDD); Treatment Resistant Depression (TRD)
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant | interventions — Ketamine; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Ketamine
  Interventions: Drug: Ketamine
- 2 (Active Comparator): Midazolam
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Ketamine — Single dose .5 mg/kg IV (in the vein) infused over 40 minutes
  Other Names: Racemic ketamine hydrochloride
  Arms: 1
Drug: Midazolam — single dose 0.045 mg/kg IV infused over 40 minutes
  Arms: 2

SUMMARY:
Existing treatments for major depressive disorder (MDD) generally take weeks to months to exert their maximal benefit. There is an urgent need to develop rapid-acting treatments for MDD. Ketamine, a high-affinity N-methyl-D-aspartate (NMDA) glutamate receptor antagonist, has been used as a standard intravenous (IV) anesthetic agent for many years in both pediatric and adult patients. Beyond its well-established role in anesthesia and pain management, there is emerging evidence that ketamine may have rapid antidepressant properties for patients with severe mood disorders.

In this study we are investigating whether ketamine can have an antidepressant effect compared to midazolam. Midazolam has similar anesthetic effects compared to ketamine but has not been shown to be an antidepressant, and is therefore acting as an active control in this study.

The study period can last up to 8 weeks, depending on your response to the study medication. There are two required overnight stays in our Research Commons as part of this study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, 21-80 years of age;
2. Female individuals who are not of childbearing potential (i.e., surgically sterile, postmenopausal for at least one year) or using a medically accepted reliable means of contraception. Women using oral contraceptive medication for birth control must also be using a barrier contraceptive. Women of childbearing potential must also have a negative serum beta-human growth hormone at screening and at pre-infusion;
3. Participants must fulfill DSM-IV criteria for Major Depression without psychotic features, based on clinical assessment by a study psychiatrist and confirmed by a structured diagnostic interview, the Structured Clinical Interview for DSM-IV TR Axis I Disorders, Patient Edition (SCID-P);
4. Participants must have a history of at least one previous episode of depression prior to the current episode (recurrent MDD) or have chronic MDD (of at least two years' duration);
5. Participants have not responded to three or more adequate trials of an antidepressant as determined by Antidepressant Treatment History Form (ATHF) criteria (score >=3);
6. Participant scores on the IDS-C30 must be greater than or equal to 32 at both Screening and within 24 hours prior to Visit 1a (Phase 1);
7. Current major depressive episode is of at least 4 weeks duration.
8. Each participant must have a level of understanding sufficient to agree to all tests and examinations required by the protocol and must sign an informed consent document;
9. Each participant must be able to identify a family member, physician, or friend who will participate in the Treatment Contract.

Exclusion Criteria:

1. Lifetime history of psychotic features, diagnosis of schizophrenia or any other psychotic disorder, or diagnosis of bipolar disorder
2. Lifetime histories of autism, mental retardation, pervasive developmental disorders, or Tourette's syndrome;
3. Current diagnosis of Obsessive Compulsive Disorder or eating disorder (bulimia nervosa or anorexia nervosa);
4. Subjects with DSM-IV drug or alcohol abuse/dependence within the preceding 2 years;
5. Patients with schizotypal or antisocial personality disorder, or any clinically significant axis II disorder that would, in the investigator's judgment, preclude safe study participation;
6. Patients judged clinically to be at serious and imminent suicidal or homicidal risk;
7. Women who are either pregnant or nursing;
8. Serious, unstable medical illnesses including hepatic, renal, gastroenterologic (including gastroesophageal reflux disease), respiratory (including obstructive sleep apnea, or history of difficulty with airway management during previous anesthetics), cardiovascular (including ischemic heart disease and uncontrolled hypertension), endocrinologic, neurologic (including history of severe head injury), immunologic, or hematologic disease;
9. Clinically significant abnormal findings of laboratory parameters, physical examination, or ECG;
10. Patients with one or more seizures without a clear and resolved etiology;
11. Patients starting hormonal treatment (e.g., estrogen) in the last 3 months prior to Visit 1a;
12. Treatment with an irreversible MAOI or any other FDA approved Anti depressant medication within one week prior to Visit 1a (with the exception of a stable dose of non-benzodiazepines hypnotics i.e. zolpidem, eszopiclone, etc for at least 3 months);
13. Treatment with fluoxetine within 4 weeks prior to Visit 1a;
14. Evidence-based individual psychotherapy (e.g. CBT or IPT) and other non-pharmacological antidepressant treatments (e.g. light therapy) will not be permitted during the acute study period (7 day);
15. Previous recreational use of PCP or Ketamine.
16. Past intolerance or hypersensitivity to midazolam
17. Hypertension (systolic BP >160 mm Hg or diastolic BP >90 mm Hg) not controlled by diuretic or beta-blocker therapy alone or in combination.
18. Evidence of age-related cognitive decline or mild dementia suggested by a score of < 27 on the Mini-Mental State Examination (MMSE) at Screening

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2008-11; Primary Completion 2012-09 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay J. Mathew, MD, Principal Investigator — Baylor College of Medicine; Dan V Iosifescu, MD,M.Sc., Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - Mount Sinai School of Medicine, New York, New York
  - Michael E. Dabakey VA Medical Center & Baylor College of Medicine, Houston, Texas

REFERENCES:
- [Background] Zarate CA Jr, Singh JB, Carlson PJ, Brutsche NE, Ameli R, Luckenbaugh DA, Charney DS, Manji HK. A randomized trial of an N-methyl-D-aspartate antagonist in treatment-resistant major depression. Arch Gen Psychiatry. 2006 Aug;63(8):856-64. doi: 10.1001/archpsyc.63.8.856. PMID 16894061
- [Background] Berman RM, Cappiello A, Anand A, Oren DA, Heninger GR, Charney DS, Krystal JH. Antidepressant effects of ketamine in depressed patients. Biol Psychiatry. 2000 Feb 15;47(4):351-4. doi: 10.1016/s0006-3223(99)00230-9. PMID 10686270
- [Derived] Wan LB, Levitch CF, Perez AM, Brallier JW, Iosifescu DV, Chang LC, Foulkes A, Mathew SJ, Charney DS, Murrough JW. Ketamine safety and tolerability in clinical trials for treatment-resistant depression. J Clin Psychiatry. 2015 Mar;76(3):247-52. doi: 10.4088/JCP.13m08852. PMID 25271445
- [Derived] Murrough JW, Iosifescu DV, Chang LC, Al Jurdi RK, Green CE, Perez AM, Iqbal S, Pillemer S, Foulkes A, Shah A, Charney DS, Mathew SJ. Antidepressant efficacy of ketamine in treatment-resistant major depression: a two-site randomized controlled trial. Am J Psychiatry. 2013 Oct;170(10):1134-42. doi: 10.1176/appi.ajp.2013.13030392. PMID 23982301

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study enrolled patients at two academic sites, Baylor College of Medicine and Icahn School of Medicine at Mount Sinai, between November 2010 and August 2012.
Pre-assignment Details: The protocol required patients to be drug free prior to the infusion, for at at least 1 week (4 for fluoxetine) for those taking other medications. Randomly assigned in a 2:1 ratio, the patients received a single intravenous infusion of ketamine hydrochloride (0.5 mg/kg) or midazolam (0.045 mg/kg) infused over 40 minutes.
Groups:
- Ketamine: single infusion of 0.5mg/kg of Ketamine HCL
- Midazolam: single infusion of midazolam being used as an active control for the study
Period: 24 Hour Endpoint
Arm/Group | Ketamine | Midazolam
Started | 48 | 25
Completed | 47 | 25
Not Completed | 1 | 0
Period: 7 Day Endpoint
Arm/Group | Ketamine | Midazolam
Started | 47 | 25
Completed | 45 | 22
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Ketamine: Ketamine
- Midazolam: Midazolam
- Total: Total of all reporting groups
Arm/Group | Ketamine | Midazolam | Total
Number analyzed (Participants) | 48 | 25 | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.9 (12.8) | 42.7 (11.6) | 44.8 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 11 | 38
  Male | 21 | 14 | 35
Region of Enrollment [Number; unit: participants]
  United States | 48 | 25 | 73

OUTCOME MEASURES:

1. Primary Outcome: MADRS
Description: Montgomery-Asberg Depression Rating Scale, each of the ten items can be scored from 0 (absence of symptoms to 6 most severe) and has a total score range of 0-60. A lower score on a MADRS indicates a less severe depression.
Time Frame: 24 hours post-infusion
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Ketamine | Midazolam
Number analyzed (Participants) | 47 | 25
units on a scale | 14.77 [11.73 to 17.80] | 22.72 [18.85 to 26.59]

ADVERSE EVENTS:
Arm/Group | Ketamine | Midazolam
Serious Adverse Events (participants affected / at risk) | 2/47 | 0/25
Other Adverse Events (participants affected / at risk) | 47/47 | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine (N=47) | Midazolam (N=25)
Hypotension/Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) — Hypotension (BP=73/40 for 1 min)/bradycardia (HR <30 bpm for 30 sec, followed by spontaneous recovery). This occurred while the subject was undergoing venipuncture at the 30 min time point and was considered a vaso- vagal episode.
Suicide Attempt (Social circumstances) | 1 (1) | 0 (0) — Suicide Attempt: While tapering off of psychotropic medication, patient was hospitalized following an attempted overdose.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ketamine (N=47) | Midazolam (N=25)
Nausea (Gastrointestinal disorders) | 16 | 3
Headache (Nervous system disorders) | 15 | 5
Dizziness on standing (Nervous system disorders) | 10 | 2
Dry Mouth (Gastrointestinal disorders) | 12 | 4
Poor Concentration (Nervous system disorders) | 19 | 12

LIMITATIONS AND CAVEATS:
Limitations of our trial include stringent enrollment criteria due to concerns about ketamine's psychoactive effects and abuse liability. A proportion of screened patients (17.2%) refused or were unable to tolerate psychotropic washout.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No